CLINICAL TRIAL: NCT04496908
Title: Early Versus Delayed Artificial Rupture of Membranes Following Foley Catheter Ripening in Labor Induction: A Randomized Controlled Trial (AROM Trial)
Brief Title: Early Versus Delayed Artificial Rupture of Membranes (AROM Trial)
Acronym: AROM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Principal Investigator, Helen Beatriz Gomez, Resident Physician, Christiana Care Health Services
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DDD# 604698
Record Dates: First submitted 2020-07-27; First posted 2020-08-04 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-11

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Amniotomy; Misoprostol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early Amniotomy (Active Comparator): Women in the Early AROM group will under amniotomy one hour from Foley Catheter expulsion. Labor augmentation will continue per study protocol. Refer to Appendix A for protocol regimen.
  Interventions: Procedure: amniotomy; Device: Foley Catheter; Drug: Misoprostol
- Delayed Amniotomy (Active Comparator): Women in the Delayed AROM group will undergo amniotomy at the discretion of the obstetrician or labor provider. No specific instructions will be given.
  Interventions: Procedure: amniotomy; Device: Foley Catheter; Drug: Misoprostol

INTERVENTIONS:
Procedure: amniotomy — Artificially rupturing membranes
Device: Foley Catheter — Foley catheter device is commonly used for cervical ripening during labor induction. It is used independently or in combination with pharmacologic augmentation. It is inserted in the cervix and the balloon is then inflated with 60 cc of saline.
Drug: Misoprostol — Misoprostol is a medication that is commonly used for cervical ripening during labor induction. It is commonly used independently or in combination with mechanical methods, such as a foley catheter. The commonly used dose during term labor induction is 25 mcg.

SUMMARY:
This randomized controlled trial of consenting women undergoing induction of labor with combined combination Foley catheter and pharmacologic cervical ripening seeks to efficacy of early amniotomy.

This project will include 157 women presenting at Christiana Care Health System. Women will be included if they are at least 37 weeks gestation, have a singleton pregnancy, have intact membranes and are undergoing an induction of labor using a Foley catheter combined with either misoprostol or pitocin. Following admission, women will be randomized into either early or delayed amniotomy

Women will be randomized with equal probability to the intervention group using block randomization stratified by party.

Prior to discharge from the hospital, baseline demographic and clinical data will be obtained via chart review

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* full term (≥37 weeks) gestations determined by routine obstetrical guidelines
* singleton gestation in cephalic presentation
* Both nulliparous and multiparous women
* Intact membranes
* Bishop score of ≤6 and cervical dilation ≤2cm

Exclusion Criteria:

* Any contraindication to a vaginal delivery or to misoprostol
* fetal demise
* Multifetal gestation
* major fetal anomaly
* prior uterine surgery, previous cesarean section
* women with HIV, hepatitis C, hepatitis B, and women with medical conditions requiring an assisted second stage
* Additional exclusion criteria were as follows: category 3 fetal heart rate tracing, hemolysis elevated liver enzymes and low platelets (HELLP) syndrome or eclampsia, growth restriction <10th percentile (based on Hadlock growth curves) with reversal of flow in umbilical artery Doppler studies, and growth restriction <5th percentile with elevated, absent, or reversal of flow in umbilical artery Doppler studies.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-05-22 (Actual); Study Completion 2021-10-18 (Actual)

PRIMARY OUTCOMES:
time to delivery | Number of hours from removal of Foley catheter to delivery of neonate; up to 72 hours.
  time to delivery (hours) defined as time from Foley Catheter expulsion to delivery regardless of mode of delivery.

SECONDARY OUTCOMES:
Cesarean delivery rate | At time of delivery
  binary; yes/no
Time to vaginal delivery | At time of delivery
  time to delivery (hours) defined as time from Foley Catheter expulsion to delivery
Maternal length of stay | through study completion, an average of 4 days
  time from admission to discharge
Indication for cesarean delivery | At time of delivery
  discrete
Chorioamnionitis | At time of delivery
  defined by the presence of maternal fever ≥100·4°f in the presence of maternal or fetal tachycardia or fundal tenderness
3rd/4th degree perineal laceration | at time of delivery
  binary; yes/no
Blood transfusion | through study completion, an average of 1 year
  binary; yes/no
Endometritis | From time of delivery to time of hospital discharge; up to 6 weeks
  binary; yes/no
Wound separation-infection | through study completion, an average of 1 year
  binary, yes/no; defined by the need for additional wound closure or the need for antibiotics
Neonatal death | through study completion, an average of 1 year
  binary, yes/no

CONTACTS AND LOCATIONS:
Locations (1):
- Christiana Care Health Systems, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wei S, Wo BL, Qi HP, Xu H, Luo ZC, Roy C, Fraser WD. Early amniotomy and early oxytocin for prevention of, or therapy for, delay in first stage spontaneous labour compared with routine care. Cochrane Database Syst Rev. 2013 Aug 7;2013(8):CD006794. doi: 10.1002/14651858.CD006794.pub4. PMID 23926074
- [Background] Macones GA, Cahill A, Stamilio DM, Odibo AO. The efficacy of early amniotomy in nulliparous labor induction: a randomized controlled trial. Am J Obstet Gynecol. 2012 Nov;207(5):403.e1-5. doi: 10.1016/j.ajog.2012.08.032. Epub 2012 Aug 24. PMID 22959833
- [Background] Levy R, Ferber A, Ben-Arie A, Paz B, Hazan Y, Blickstein I, Hagay ZJ. A randomised comparison of early versus late amniotomy following cervical ripening with a Foley catheter. BJOG. 2002 Feb;109(2):168-72. doi: 10.1111/j.1471-0528.2002.01137.x. PMID 11888099
- [Background] Levine LD, Downes KL, Elovitz MA, Parry S, Sammel MD, Srinivas SK. Mechanical and Pharmacologic Methods of Labor Induction: A Randomized Controlled Trial. Obstet Gynecol. 2016 Dec;128(6):1357-1364. doi: 10.1097/AOG.0000000000001778. PMID 27824758
- [Background] Delaney S, Shaffer BL, Cheng YW, Vargas J, Sparks TN, Paul K, Caughey AB. Labor induction with a Foley balloon inflated to 30 mL compared with 60 mL: a randomized controlled trial. Obstet Gynecol. 2010 Jun;115(6):1239-1245. doi: 10.1097/AOG.0b013e3181dec6d0. PMID 20502296
- [Derived] Gomez Slagle HB, Fonge YN, Caplan R, Pfeuti CK, Sciscione AC, Hoffman MK. Early vs expectant artificial rupture of membranes following Foley catheter ripening: a randomized controlled trial. Am J Obstet Gynecol. 2022 May;226(5):724.e1-724.e9. doi: 10.1016/j.ajog.2021.11.1368. Epub 2022 Feb 6. PMID 35135684